CLINICAL TRIAL: NCT07131722
Title: An Open-Label, Dose-Finding, Phase 1/2a Study to Evaluate the Efficacy and Safety of PRG-N-01 in Patients With Neurofibromatosis Type II
Brief Title: Study to Determine Optimal Dose, Evaluate the Efficacy and Safety of PRG-N-01 in Patients With Neurofibromatosis Type II
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: PRG Science & Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PRG-NF-001
Record Dates: First submitted 2025-07-01; First posted 2025-08-20 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-08

CONDITIONS: Neurofibromatosis Type II; NF2
MeSH Terms: conditions — Neurofibromatosis 2

STUDY DESIGN:
Intervention Model Description: Sequential Assignment, non-Randomized (Phase 1), then Parallel Assignment, Randomized (Phase 2a)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Trineumin Dose Escalation Arm (Experimental): Subjects receive Trineumin(Code: name: PRG-N-01) orally once daily across six sequential dose cohorts. Dose escalation follows an accelerated titration design (Cohort 1), a 3+3 design (Cohort 2), and a rolling 6 design thereafter. Dosing proceeds unless dose-limiting toxicities (DLTs) are observed.
  Interventions: Drug: Trineumin
- Trineumin Low Dose (Phase 2a) (Experimental): Subjects receive Trineumin(Code: name: PRG-N-01) at the selected lower dose (e.g., RP2D or sub-RP2D level) once daily. Subjects are randomized in Phase 2a.
  Interventions: Drug: Trineumin
- Trineumin High Dose (Phase 2a) (Experimental): Subjects receive Trineumin(Code: name: PRG-N-01) at a higher dose once daily in Phase 2a. Subjects are randomized to this arm.
  Interventions: Drug: Trineumin

INTERVENTIONS:
Drug: Trineumin — Trineumin(Code name: PRG-N-01) is administered orally once daily. The study includes six dose levels.
  Dose escalation decisions are based on observed DLTs.
  Arms: Trineumin Dose Escalation Arm
Drug: Trineumin — Trineumin(Code name: PRG-N-01) is administered orally once daily at the lower dose selected from Phase 1 results.
  Arms: Trineumin Low Dose (Phase 2a)
Drug: Trineumin — Trineumin(Code name: PRG-N-01) is administered orally once daily at the higher dose selected from Phase 1 results.
  Arms: Trineumin High Dose (Phase 2a)

SUMMARY:
The goal of this clinical trial is to learn if Trineumin(Code name:PRG-N-01) works to treat Neurofibromatosis Type II(NF2) in adults. It will also learn about the safety and tolerability and toxicity of PRG-N-01. The main questions it aims to answer are:

* What dose was determined as the Maximum Tolerated Dose (MTD) of Trineumin?
* What dose was explored as the optimal effective dose of Trineumin based on radiographic response?
* Does Trineumin reduce tumor size or improve participants' quality of life, including hearing function?
* What medical problems do participants have when taking Trineumin?

Participants will:

* Take Trineumin every day for 96 weeks
* Visit the clinic once 1, 4, 8, 12, 18week and every 12 weeks and for checkups and tests

DETAILED DESCRIPTION:
This is an open-label, Phase 1/2a clinical study to evaluate the safety, tolerability, pharmacokinetics, and preliminary efficacy of Trineumin(Code name:PRG-N-01) in subjects with Neurofibromatosis Type II(NF2)-related tumors

Phase 1 Subjects who voluntarily provide written informed consent will be screened according to predefined inclusion and exclusion criteria. The Phase 1 portion is designed to determine the maximum tolerated dose (MTD) and recommended Phase 2 dose (RP2D) of Trineumin.

A total of six dose levels are planned. Dose escalation follows an accelerated titration design (ATD) for Cohort 1, a standard 3+3 design for Cohort 2, and a rolling six design for subsequent cohorts. Trineumin is administered orally once daily. Each subject is assigned to a cohort in the order of enrollment. The dose-limiting toxicity (DLT) observation period is 12 weeks following initial dosing. Subjects without DLT or who recover from DLT during this period may continue treatment.

Phase 2a In the Phase 2a portion, eligible subjects who provide informed consent will be randomized to receive one of two selected doses of Trineumin orally once daily. Randomization is stratified based on predefined criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged 18 years or older at screening
2. Subjects diagnosed with NF2 clinically or genetically, according to the I-NF-DC 2022 updated NF2 diagnostic criteria
3. Subjects with tumors due to NF2 who require treatment if they meet one of more of the criteria below but cannot undergo surgical treatment due to high risk of side effects from surgery (e.g., damage to nerve function).

(1) Subjects with progressive tumors (VS, non-VS, meningiomas, ependymomas) confirmed on MRI within 36 months prior to screening (2) Subjects with clinical symptoms (decreased function of affected nerves, such as hearing loss, uncontrolled pain, shortness of breath, difficulty swallowing, decreased motor function, and decreased gait) as judged by the investigator 4) Subjects with ECOG performance status 0 - 1 or Karnofsky performance status 70 or higher 5) Subjects who have appropriate hematological, liver, renal, and blood coagulation functions confirmed based on the following criteria at screening: 6) Subjects who have appropriate cardiac and pulmonary functions confirmed based on the following criteria at screening: 7) Subjects who agree to use sunscreen during the clinical study period. 8) Subjects (or the subject's legal representative) who voluntarily consent and provide written informed consent to participate in this clinical study.

9) (Only for Phase 2a) Subjects with one or more measurable NF2-related tumors confirmed on MRI at screening

Exclusion Criteria:

1) Subjects who have the following past or current medical history confirmed during screening:

(1) Malignant tumor requiring treatment (chemotherapy or radiotherapy) or with disease progression within 2 years prior to screening (2) The following heart-related history

* Uncontrolled hypertension at screening (DBP ≥100 mmHg or SBP ≥160 mmHg despite treatment)
* Acute coronary syndrome (ACS) within 24 weeks of baseline, clinically significant arrhythmia, cardiomyopathy, unstable angina, NYHA II-IV heart failure, or severe valvular heart disease

  1. Interstitial lung disease or pulmonary fibrosis
  2. Cystitis or urinary obstruction within 12 weeks prior to screening
  3. Blood coagulation disorder
  4. Severe or active infectious disease requiring antibiotics, antivirals, etc. within 4 weeks prior to screening
  5. Gastrointestinal disease that currently makes oral administration difficult or may affect absorption (e.g., celiac disease, Crohn's disease, intestinal resection)
  6. Other diseases that are sufficient to affect the clinical study results at the investigator's discretion.

  2) Subjects who have confirmed or need the following drug treatments:
  1. Chemotherapy, immunotherapy, or myelosuppressive chemotherapy within 4 weeks prior to screening (but, within 6 weeks prior to screening for nitrosourea agents or mitomycin C)
  2. Monoclonal antibody therapy within 12 weeks prior to screening (but, allowing if more than 3 half-lives have elapsed); stem cell transplantation (but, allowing if there is no evidence of active graft-versus-host disease and more than 12 weeks have elapsed since transplantation)
  3. Other investigational drugs or devices within 4 weeks prior to screening
  4. Corticosteroids such as prednisone and prednisolone within 1 week prior to screening (but, allowing if treated with low doses)
  5. Substrate of strong inhibitor, inducer, or transporter (OCT2, MATE1, MATE2-K) of CYP enzymes (CYP2C8, CYP3A) (but, allowing only if more than 5 times the half-life from baseline has elapsed) 3) Subjects who performed a major surgery within 4 weeks prior to screening (but, allowing minor surgical procedures such as catheter replacement therapy and local biopsy).

  4) Subjects who received radiation therapy for the purpose of treating tumors due to NF2 within 24 weeks prior to screening or who require total body irradiation during the clinical study period.

  5) Subjects with prosthetics or orthopedic devices that may interfere with the volumetric analysis of target lesions via MRI.

  6) Subjects with a known severe hypersensitivity to PRG-N-01 or a concomitant medication or the ingredients or a history of allergic reactions to compounds of similar chemical or biological composition.

  7) Female subjects who are pregnant or breastfeeding 8) Women of childbearing potential or men who are unwilling to use an appropriate method of contraception from the date of written consent to 12 weeks after the last dose of PRG-N-01.

  9) Other subjects who are deemed unsuitable for participation in this clinical study at the investigator's discretion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2026-07 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Phase 1_Incidence of Dose-Limiting Toxicities (DLTs) | Each treatment group at the 12-week time point after IP administration
  Incidence of DLTs will be assessed to determine the MTD and RP2D based on predefined criteria.
Phase 1_Maximum Tolerated Dose (MTD) | Each treatment group at the 12-week time point after IP administration
  it determine the MTD based on predefined criteria.
Phase 1_ Recommended Phase 2 Dose (RP2D) | Each treatment group at the 12-week time point after IP administration
  it determine the RP2D based on predefined criteria.
Phase2a_Maximum tumor size change rate of Radiographic Tumor Response | From baseline excluding week 24 to week 96 at 12-week intervals
  Based on best overall response (BOR), ORR, DOR, PFS, and changes in tumor size from baseline using up to 4 target lesions.
Phase2a_best overall response (BOR) of Radiographic Tumor Response | From baseline excluding week 24 to week 96 at 12-week intervals
  Based on best overall response (BOR), ORR, DOR, PFS, and changes in tumor size from baseline using up to 4 target lesions.
Phase2a_Objective response rate (ORR) of Radiographic Tumor Response | From baseline excluding week 24 to week 96 at 12-week intervals
  Based on best overall response (BOR), ORR, DOR, PFS, and changes in tumor size from baseline using up to 4 target lesions.
Phase2a_Duration of response (DOR) of Radiographic Tumor Response | From baseline excluding week 24 to week 96 at 12-week intervals
  Based on best overall response (BOR), ORR, DOR, PFS, and changes in tumor size from baseline using up to 4 target lesions.
Phase2a_Progression-free survival (PFS) of Radiographic Tumor Response | From baseline excluding week 24 to week 96 at 12-week intervals
  Based on best overall response (BOR), ORR, DOR, PFS, and changes in tumor size from baseline using up to 4 target lesions.

SECONDARY OUTCOMES:
Phase1_Progression-free survival (PFS) of Radiographic Tumor Response | From baseline to week 96 at 12-week intervals
Phase1_Duration of response (DOR) of Radiographic Tumor Response | From baseline to week 96 at 12-week intervals
Phase1_Objective response rate (ORR) of Radiographic Tumor Response | From baseline to week 96 at 12-week intervals
Phase1_best overall response (BOR) of Radiographic Tumor Response | From baseline to week 96 at 12-week intervals
Phase1_Maximum tumor size change rate of Radiographic Tumor Response | From baseline to week 96 at 12-week intervals
Phase1,2a_ Pure Tone Audiometry (PTA) in Functional Hearing Response | From baseline to week 96 at 12-week intervals
Phase1,2a_Word Recognition Score (WRS) in Functional Hearing Response | From baseline to week 96 at 12-week intervals
Phase1,2a_Change of NFTI-QOL scores in Quality of Life | From baseline to week 96 at 12-week intervals
Phase1,2a_Change of PAN-QOL scores in Quality of Life | From baseline to week 96 at 12-week intervals
Phase1,2a_Incidence and Severity of Adverse Events | Up to 108 weeks
  adverse events will be recorded and graded according to CTCAE v5.0

OTHER OUTCOMES:
Phase2a_ Exploratory Analysis of Biomarker Expression in Blood | Day 1,Week 12,Week 36
  Blood samples will be collected and stored during Phase 2a for exploratory analysis of biomarkers.
Phase 1,2a_ AUC last of Day1 | Day 1, Day 7, and At every visit until week 96
Phase 1,2a_ AUCinf of Day1 | Day 1, Day 7, and At every visit until week 96
Phase 1,2a_ Cmax of Day1 | Day 1, Day 7, and At every visit until week 96
Phase 1,2a_ Tmax of Day1 | Day 1, Day 7, and At every visit until week 96
Phase 1,2a_ CL/F of Day1 | Day 1, Day 7, and At every visit until week 96
Phase 1,2a_ Vd/F of Day1 | Day 1, Day 7, and At every visit until week 96
Phase 1,2a_ t1/2 of Day1 | Day 1, Day 7, and At every visit until week 96
Phase 1,2a_ AUCtau,ss of Day 7 | Day 1, Day 7, and At every visit until week 96
Phase 1,2a_ Cmax,ss of Day 7 | Day 1, Day 7, and At every visit until week 96
Phase 1,2a_ Cmin,ss of Day 7 | Day 1, Day 7, and At every visit until week 96
Phase 1,2a_ Cav,ss of Day 7 | Day 1, Day 7, and At every visit until week 96
Phase 1,2a_ PTF (Peak-trough fluctuation) of Day 7 | Day 1, Day 7, and At every visit until week 96
Phase 1,2a_ Tmax,ss of Day 7 | Day 1, Day 7, and At every visit until week 96
Phase 1,2a_ CLss/F of Day 7 | Day 1, Day 7, and At every visit until week 96
Phase 1,2a_ Vdss/F of Day 7 | Day 1, Day 7, and At every visit until week 96
Phase 1,2a_t1/2,ss of Day 7 | Day 1, Day 7, and At every visit until week 96
Phase 1,2a_ Accumulation ratio of Day 7 | Day 1, Day 7, and At every visit until week 96